CLINICAL TRIAL: NCT02104544
Title: Investigation of DHA Intake in Pregnant and Lactating Women in China
Status: Completed | Type: Observational
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Liu Jianmeng, The Institute of Reproductive and Child Health, Peking University
Other Study IDs: 14.10.CN.INF
Record Dates: First submitted 2014-04-01; First posted 2014-04-04 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Nutrient Intake Disorder
Keywords: DHA intake;; Plasma;; Erythrocyte;; Breast milk.

STUDY DESIGN:
Observational Model: Cohort
Biospecimen Retention: Samples Without DNA — 1. Collection of venous blood, pretreatment of blood sample, take the plasma and erythrocyte respectively.
  2. Collection of breast milk (only for women having lactated for 42±7 days)
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is a multi-center, cross-sectional, non-interventional, observational study--an investigation carried out in 816 pregnant (pregnant week 17±2 group and pregnant week 39±2 group; 408 cases in each group) and 408 lactating women (post-natal lactation day 42±7 group) from a total of 4 sites in 3 typical areas (1 coastal regions, 2 inland regions and 1 lake regions) in China to study the correlation between DHA intake and DHA concentrations in blood and breast milk.

DETAILED DESCRIPTION:
This is a multi-center, cross-sectional, non-interventional, observational study in 816 pregnant (gestation week 17±2 group and gestation week 39±2 group 408 cases in each group) and 408 lactating women (post-natal lactation day 42±7 group) from a total of 4 sites in 3 typical areas (1 coastal regions, 2 inland regions and 1 lake regions) in China to study the correlation between DHA intake and DHA concentrations in blood and breast milk. Investigators are mainly physicians majoring in gynaecology and obstetrics, etc. During visits, the study physician will record the patient's social demographic data, disease and relevant medication history, review her medical records, assess DHA intake by the DHA Screener, and determine DHA concentrations in erythrocyte membrane, plasma and breast milk, so as to validate the feasibility of DHA Screener as DHA intake assessment tool for determining DHA concentrations in the body.

Subjects meeting inclusion criteria and non of the exclusion criteria will be informed of relevant information of the study. Subjects should be voluntarily consent to participate in the study and sign the informed consent form.

Screening of the study is scheduled for as long as 5 months. In this study, additional examinations or other interventions are not required.

ELIGIBILITY:
Inclusion Criteria:

PREGNANT WOMEN:

* Healthy women presenting at their week 17±2 and week 39±2 obstetric examination;
* 18-40 years of age;
* Monocyesis;
* Having signed the informed consent form voluntarity before participating in the study.

LACTATING WOMEN:

* Healthy women presenting at their day 42±7 post-natal visit;
* 18-40 years of age;
* Monocyesis;
* Having signed the informed consent form voluntarily before participating in the study

Exclusion Criteria:

* Administration of DHA supplements (milk powder for pregnant women, DHA soft capsule, Zmarto, NURIZ, Naturies, HeadDHA, Beibeicong, Nutrimed etc);
* Still experiencing severe vomiting after 16 weeks of pregnancy;
* Women who have heart, liver, kidney, (ALT and AST≥ 1.5 times of normal upper limit, Cr>normal upper limit) or severe lung disease or laboratory abnormality (i.e.lipid metabolism disorder) that may interfere with the interpretation of study results, as indicated in previous examinations;
* Pregnant woman currently participating in other clinical trials or who have participated in another clinical trial in the last 30 days;
* Women who in the judgement of the investigator cannot be expected to comply with the protocol or study procedures.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 816 pregnant (pregnant week 17±2 group and pregnant week 39±2 group; 408 cases in each group) and 408 lactating women (post-natal lactation day 42±7 group)
Sampling Method: Non-Probability Sample
Enrollment: 1254 (Actual)
Dates: Start 2014-04; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
To evaluate the feasibility in using DHA Screener for determination of internal DHA concentration | 5 months
  Correlation between DHA Screener and DHA concentration in plasma; Correlation between DHA Screener and DHA concentration in erythrocyte membrane; Correlation between DHA Screener and DHA concentration in breast milk.

SECONDARY OUTCOMES:
To compare the correlation between DHA Screener and RBC DHA among different subgroups. To compare DHA intake assessed by DHA Screener against Chinese recommendations of DHA intake. | 5 months
  1. To assess correlation between DHA Screener assessment tool and RBC DHA among study groups;
  2. To compare DHA intake assessed by DHA Screener against Chinese recommendations of DHA intake.
To compare DHA intake assessed by DHA Screener against Chinese recommendations of DHA intake. | 5 months
  To compare DHA intake assessed by DHA Screener against Chinese recommendations of DHA intake.

OTHER OUTCOMES:
To assess the correlation between DHA intake and DHA concentrations in the blood and breast milk of lactating women | 5 months
  To assess the correlation between DHA intake and DHA concentrations in the blood and breast milk of lactating women

CONTACTS AND LOCATIONS:
Overall Officials: Jianmeng Liu, Doctor, Study Chair — Peking University